CLINICAL TRIAL: NCT01254396
Title: An Open Label Crossover Study In Healthy Older Male Subjects To Evaluate The Pharmacokinetics And Safety Of An Orally Disintegrating Tablet Formulation Of Sildenafil Administered Without Water Under Fed Compared To Fasted Conditions
Brief Title: Pharmacokinetics Of Sildenafil Orally Disintegrating Tablet Formulation Given With Or Without Food.
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer's Upjohn has merged with Mylan to form Viatris Inc. (Industry)
Responsible Party: Sponsor
Organization: Pfizer (Industry)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: A1481290
Record Dates: First submitted 2010-11-19; First posted 2010-12-06 (Estimated); Results first posted 2012-02-08 (Estimated); Last update posted 2021-02-01 (Actual); Status verified 2021-01

CONDITIONS: Erectile Dysfunction
Keywords: Bioavailability Food Effect Oral Dissolving Tablet (ODT)
MeSH Terms: conditions — Erectile Dysfunction | interventions — Sildenafil Citrate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Sildenafil ODT tablet 50 mg, Fasted (Active Comparator): Treatment A: Sildenafil ODT tablet 50 mg, administered without water under fasted conditions.
  Interventions: Drug: Sildenafil
- Sildenafil ODT tablet 50 mg, Fed (Experimental): Treatment B: Sildenafil ODT tablet 50 mg, administered without water under fed conditions.
  Interventions: Drug: Sildenafil

INTERVENTIONS:
Drug: Sildenafil — Orally Disintegrating Tablet, 50 mg, Single Dose
  Arms: Sildenafil ODT tablet 50 mg, Fasted
Drug: Sildenafil — Orally Disintegrating Tablet, 50 mg, Single Dose
  Arms: Sildenafil ODT tablet 50 mg, Fed

SUMMARY:
This study will evaluate if an orally disintegrating tablet of sildenafil will have similar pharmacokinetic properties when given with food and without food.

ELIGIBILITY:
Inclusion Criteria:

* Otherwise healthy male subjects age 45 years or older with or without erectile dysfunction.
* Body Mass Index (BMI) of 17.5 to 32.5 kg/m2.
* Signed Informed Consent.

Exclusion Criteria:

* Evidence or history of clinically significant abnormalities
* Have baseline orthostatic hypotension
* Positive drug screen, excessive alcohol and tobacco use

Min Age: 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2010-12; Primary Completion 2011-01 (Actual); Study Completion 2011-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer Investigational Site, Singapore, Singapore

REFERENCES:
- [Derived] Damle B, Duczynski G, Jeffers BW, Crownover P, Coupe A, LaBadie RR. Pharmacokinetics of a novel orodispersible tablet of sildenafil in healthy subjects. Clin Ther. 2014 Feb 1;36(2):236-44. doi: 10.1016/j.clinthera.2013.12.010. Epub 2014 Jan 18. PMID 24447534
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A1481290&StudyName=Pharmacokinetics%20Of%20Sildenafil%20Orally%20Disintegrating%20Tablet%20Formulation%0AGiven%20With%20Or%20Without%20Food.%20%20%0A

RESULTS

PARTICIPANT FLOW:
Groups:
- Sildenafil Fasted First, Then Sildenafil Fed: Single oral dose of sildenafil 50 milligram (mg) orally disintegrating tablet (ODT) under fasted condition in first intervention period; and single oral dose of sildenafil 50 mg ODT under fed condition in second intervention period. A washout period of at least 1 day was maintained between each period.
- Sildenafil Fed First, Then Sildenafil Fasted: Single oral dose of sildenafil 50 mg ODT under fed condition in first intervention period; and single oral dose of sildenafil 50 mg ODT under fasted condition in second intervention period. A washout period of at least 1 day was maintained between each period.
Period: First Intervention Period
Arm/Group | Sildenafil Fasted First, Then Sildenafil Fed | Sildenafil Fed First, Then Sildenafil Fasted
Started | 6 | 6
Completed | 6 | 6
Not Completed | 0 | 0
Period: Washout Period (at Least 1 Day)
Arm/Group | Sildenafil Fasted First, Then Sildenafil Fed | Sildenafil Fed First, Then Sildenafil Fasted
Started | 6 | 6
Completed | 6 | 6
Not Completed | 0 | 0
Period: Second Intervention Period
Arm/Group | Sildenafil Fasted First, Then Sildenafil Fed | Sildenafil Fed First, Then Sildenafil Fasted
Started | 6 | 6
Completed | 6 | 6
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Entire Study Population: Includes groups randomized to receive sildenafil 50 mg ODT under fasted condition first and sildenafil 50 mg ODT under fed condition first.
Arm/Group | Entire Study Population
Number analyzed (Participants) | 12
Age, Continuous [Mean (Standard Deviation); unit: years] | 56.6 (8.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 12

OUTCOME MEASURES:

1. Primary Outcome: Maximum Observed Plasma Concentration (Cmax)
Time Frame: 0 (pre-dose), 0.25, 0.5, 0.75, 1, 1.5, 2, 3, 4, 6, 8, 10, 12 and 14 hrs post-dose
Population: Pharmacokinetic parameter analysis population included all randomized and treated participants who had at least 1 of the pharmacokinetic parameters of primary interest in at least 1 treatment period.
Measure: Geometric Mean (Standard Deviation); unit: ng/mL
Groups:
- Sildenafil 50 mg (Fasted): Single oral dose of sildenafil 50 mg ODT under fasted condition (Reference) in either first intervention period or second intervention period.
- Sildenafil 50 mg (Fed): Single oral dose of sildenafil 50 mg ODT under fed condition (Test) in either first intervention period or second intervention period.
Arm/Group | Sildenafil 50 mg (Fasted) | Sildenafil 50 mg (Fed)
Number analyzed (Participants) | 12 | 12
ng/mL | 292.60 (93.84) | 121.00 (56.92)
Statistical Analysis 1: Comparison: Sildenafil 50 mg (Fasted) vs Sildenafil 50 mg (Fed); Natural log transformed Cmax of sildenafil was analyzed using a mixed effect model with sequence, period and treatment as fixed effects and participant within sequence as a random effect. The adjusted mean differences and 90% confidence intervals for the differences were exponentiated to provide estimates of the ratio of adjusted geometric means (Test/Reference) and 90% confidence intervals for the ratios; Test type: Superiority or Other; Ratio of Adjusted Means = 41.35, 90% CI 2-sided [32.40 to 52.76]

2. Secondary Outcome: Time to Reach Maximum Observed Plasma Concentration (Tmax)
Time Frame: 0 (pre-dose), 0.25, 0.5, 0.75, 1, 1.5, 2, 3, 4, 6, 8, 10, 12 and 14 hrs post-dose
Population: as for outcome 1
Measure: Median (Full Range); unit: hrs
Arm/Group | Sildenafil 50 mg (Fasted) | Sildenafil 50 mg (Fed)
Number analyzed (Participants) | 12 | 12
hrs | 0.625 [0.250 to 1.500] | 4.000 [0.500 to 6.000]

3. Secondary Outcome: Area Under the Curve From Time Zero to Extrapolated Infinite Time [AUC (0-∞)]
Description: AUC (0-∞) = Area under the plasma concentration versus time curve (AUC) from time zero (pre-dose) to extrapolated infinite time (0-∞). It is obtained from AUC (0-t) plus AUC (t-∞).
Time Frame: 0 (pre-dose), 0.25, 0.5, 0.75, 1, 1.5, 2, 3, 4, 6, 8, 10, 12 and 14 hrs post-dose
Population: Pharmacokinetic parameter analysis population included all randomized and treated participants who had at least 1 of the pharmacokinetic parameters of primary interest in at least 1 treatment period. Here, the 'N' (number of participants analyzed) is signifying those participants who were evaluable for this measure.
Measure: Geometric Mean (Standard Deviation); unit: ng*hr/mL
Arm/Group | Sildenafil 50 mg (Fasted) | Sildenafil 50 mg (Fed)
Number analyzed (Participants) | 12 | 9
ng*hr/mL | 838.60 (197.20) | 804.00 (284.69)
Statistical Analysis 1: Comparison: Sildenafil 50 mg (Fasted) vs Sildenafil 50 mg (Fed); Natural log transformed AUC (0-∞) of sildenafil was analyzed using a mixed effect model with sequence, period and treatment as fixed effects and participant within sequence as a random effect. The adjusted mean differences and 90% confidence intervals for the differences were exponentiated to provide estimates of the ratio of adjusted geometric means (Test/Reference) and 90% confidence intervals for the ratios; Test type: Superiority or Other; Ratio of Adjusted Means = 93.42, 90% CI 2-sided [80.23 to 108.78]

4. Primary Outcome: Area Under the Curve From Time Zero to Last Quantifiable Concentration (AUClast)
Description: Area under the plasma concentration time-curve from zero (pre-dose) to the last measured concentration (AUClast).
Time Frame: 0 (pre-dose), 0.25, 0.5, 0.75, 1, 1.5, 2, 3, 4, 6, 8, 10, 12 and 14 hours (hrs) post-dose
Population: as for outcome 1
Measure: Geometric Mean (Standard Deviation); unit: ng*hr/mL
Arm/Group | Sildenafil 50 mg (Fasted) | Sildenafil 50 mg (Fed)
Number analyzed (Participants) | 12 | 12
ng*hr/mL | 813.20 (186.29) | 712.80 (245.58)
Statistical Analysis 1: Comparison: Sildenafil 50 mg (Fasted) vs Sildenafil 50 mg (Fed); Natural log transformed AUClast of sildenafil was analyzed using a mixed effect model with sequence, period and treatment as fixed effects and participant within sequence as a random effect. The adjusted mean differences and 90% confidence intervals for the differences were exponentiated to provide estimates of the ratio of adjusted geometric means (Test/Reference) and 90% confidence intervals for the ratios; Test type: Superiority or Other; Ratio of Adjusted Means = 87.66, 90% CI 2-sided [77.62 to 98.99]

5. Secondary Outcome: Plasma Decay Half Life (t1/2)
Description: Plasma decay half-life is the time measured for the plasma concentration to decrease by one half.
Time Frame: 0 (pre-dose), 0.25, 0.5, 0.75, 1, 1.5, 2, 3, 4, 6, 8, 10, 12 and 14 hrs post-dose
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: hrs
Arm/Group | Sildenafil 50 mg (Fasted) | Sildenafil 50 mg (Fed)
Number analyzed (Participants) | 12 | 9
hrs | 3.039 (0.484) | 2.503 (0.359)

ADVERSE EVENTS:
Description: The same event may appear as both an AE and a SAE. However, what is presented are distinct events. An event may be categorized as serious in one subject and as nonserious in another subject, or one subject may have experienced both a serious and nonserious event during the study.
Arm/Group | Sildenafil 50 mg (Fasted) | Sildenafil 50 mg (Fed)
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/12
Other Adverse Events (participants affected / at risk) | 3/12 | 3/12
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Sildenafil 50 mg (Fasted) (N=12) | Sildenafil 50 mg (Fed) (N=12)
Catheter site haematoma (General disorders) | 2 | 0
Headache (Nervous system disorders) | 0 | 1
Dry throat (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 2
Dry skin (Skin and subcutaneous tissue disorders) | 1 | 1

LIMITATIONS AND CAVEATS:
AUC (0-t) was the intended primary outcome measure.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.